CLINICAL TRIAL: NCT01475227
Title: A Randomized Crossover Study of the Effects of Zinc Sulphate Supplementation on Atazanavir/Ritonavir-associated Hyperbilirubinemia
Brief Title: Atazanavir/Ritonavir and Zinc Pharmacokinetic Study
Acronym: SSAT043
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SSAT 043
Record Dates: First submitted 2011-10-31; First posted 2011-11-21 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: HIV Infection
Keywords: HIV; Bilirubin
MeSH Terms: conditions — HIV Infections | interventions — Zinc Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A- early Solvazinc group (Experimental): Zinc sulphate 125mg (1 Solvazinc tablet) once daily orally after dissolution in water, day 2 to day 15
  Interventions: Drug: 1 Solvazinc tablet, day 2 to day 15
- Arm B- late Solvazinc group (Experimental): Zinc sulphate 125mg (1 Solvazinc tablet) once daily orally after dissolution in water, day 15 to day 28
  Interventions: Drug: 1 Solvazinc tablet, day 15 to day 28

INTERVENTIONS:
Drug: 1 Solvazinc tablet, day 2 to day 15 — Zinc sulphate 125mg, day 2 to day 15
  Other Names: Zinc sulphate
  Arms: Arm A- early Solvazinc group
Drug: 1 Solvazinc tablet, day 15 to day 28 — Zinc sulphate 125mg, day 15 to day 28
  Other Names: Zinc sulphate
  Arms: Arm B- late Solvazinc group

SUMMARY:
The study is being conducted as the most common side effect of the HIV drug atazanavir (taken with ritonavir) is hyperbilirubinaemia. Bilirubin is a normal waste product from the body and gets broken down in the liver so it can leave the body through the gut. Atazanavir slows the breakdown of this chemical, which can cause jaundice (yellowing of the skin) and/or scleral icterus (yellowing of the eyes). This is completely harmless; in fact up to 1 in 10 of the UK population have an inherited condition that causes the same yellowing. However, some patients don't like this side effect and it is the commonest reason for switching off the drug.

A study in people with Gilberts syndrome (the inherited condition that causes the same changes in the chemical bilirubin) showed that a mineral supplement (zinc sulphate) reduced the levels of bilirubin in the blood. The aim of this study is to see if using zinc supplements can achieve the same effect in patients with high bilirubin due to atazanavir use.

DETAILED DESCRIPTION:
Atazanavir is a protease inhibitor (PI) and, like other agents in this class, requires pharmacological 'boosting' with the cytochrome p450 inhibitor ritonavir. Ritonavir slows the hepatic clearance of PIs, increasing plasma concentration and allowing the us eof lower, and less frequent doses. Atazanavir, boosted with ritonavir, is approved for once-daily use, is an internationally preferred first-line agent (in combination with a backbone of two nucleosides [NRTI]) and the most commonly prescribed PI in the UK. Once-daily atazanavir/ritonavir with two NRTI is an effective and well-tolerated therapeutic option for people living with HIV infection. The most common adverse event associated with atazanavir use is unconjugated hyperbilirubinaemia. This is observed in over 40% of patients and up to 5% of patients discontinue the drug due jaundice and/or scleral icterus.

Truvada is a fixed dose combination of two NRTI, tenofovir (245mg) and emtricitabine (200mg), administered as one tablet once daily. Truvada is a preferred NRTI backbone in national and international guidelines and the first line, therefore most commonly used, NRTI backbone in our unit.

Benefits of atazanavir/ritonavir compared with alternative agents include once daily dosing, low pill burden, low rates of gastro-intestinal toxicity and, importantly in a patient population already at an elevated risk of cardiovascular disease, a favourable lipid profile. If a simple intervention could reduce the incidence of hyperbilirubinaemia this could reduce the risk of treatment discontinuation/switch. The aim of this study is to explore the benefit, and safety, of adding zinc sulphate in patients on a stable regimen of Truvada, atazanavir and ritonavir.

ELIGIBILITY:
Inclusion Criteria:

1. The ability to understand and sign a written informed consent form, prior to participation in any screening procedure and must be willing to comply with all study requirements
2. Male or non-pregnant, non-lactating females.
3. Aged between 18 to 65 years, inclusive.
4. Documented HIV-1 infection
5. Plasma HIV RNA less than 40 copies/mL (note retesting of screening viral load is allowed).
6. CD4 count > 100 at screening (note retesting of screening CD4 count is allowed).
7. Receiving an antiretroviral regimen of Truvada and atazanavir/ritonavir for more than 3 months.
8. Serum total bilirubin concentration greater than 25 micromol/L
9. Agrees not to change regimen, outside the study recommendations, from baseline until end of the treatment period unless this is medically indicated as decided by their treating physician.

Exclusion Criteria:

1. Any serious or active medical or psychiatric illness, which, in the opinion of the investigator, would interfere with subject treatment, assessment, or compliance with the protocol. This would include any active clinically significant renal, cardiac, hepatic, pulmonary, vascular, metabolic disorders or malignancy.
2. Body mass index (BMI) >35 kg/m2
3. Presence of any current active AIDS defining illness (Category C conditions according to the CDC Classification System for HIV Infection 1993) with the following exceptions:

   • Stable cutaneous Kaposi's Sarcoma
4. Clinically relevant alcohol or drug use (positive urine drug screen, with the exception of cannabinoids) or history of alcohol or drug use considered by the Investigator to be sufficient to hinder compliance with treatment, follow-up procedures or evaluation of adverse events.
5. The use of zinc supplements for 1 month before screening and disallowed concomitant therapy (See Concomitant Medication and treatment, section 5.2) or medication that may interfere with the study results (as determined by the principal investigator).
6. Females of childbearing potential who are not using effective non-hormonal birth control methods or not willing to continue using these birth control methods for at least 14 days after the end of the treatment period.
7. Previous allergy to any of the constituents of the zinc sulphate tablets administered in this trial.
8. Subjects with laboratory evidence of significantly decreased hepatic or renal function (as determined by the principal investigator).
9. Exposure to any investigational drug or placebo within 4 weeks of first dose of study drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To assess the change in unconjugated hyperbilirubinaemia following acute and chronic administration of zinc sulphate during atazanavir/ritonavir therapy. | baseline and day 29
  Change in serum unconjugated bilirubin concentrations when atazanavir/ritonavir is added to zinc sulphate, adjusted for period effect

SECONDARY OUTCOMES:
safety and tolerability of zinc sulphate supplement when given concomitantly with atazanavir/ritonavir | baseline and day 14
  Assessment of the impact of adding zinc sulphate to atazanavir/ritonavir-based HAART on grade 2-4 laboratory abnormalities and adverse events.
To assess atazanavir plasma exposure in the presence of zinc and relationship between the latter and hyperbilirubin during zinc intake. | baseline and day 14
  Atazanavir plasma exposure in the presence of zinc and relationship between the latter and hyperbilirubin during zinc intake.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, Dr, Principal Investigator — St Stephen's AIDS Trust
Locations (1):
- St Stephen's AIDS Trust, London, United Kingdom